CLINICAL TRIAL: NCT06188455
Title: Clinical Study of Fluzopalil Combined With Apatinib for Maintenance Therapy After Platinum-containing Chemotherapy in Patients With Recurrent Ovarian Cancer
Brief Title: Maintenance Therapy After Platinum-containing Chemotherapy in Patients With Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-OC-021
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fuzuloparib With Apatinib Mesylate Tablets (Experimental)
  Interventions: Drug: Fluzoparib Capsules; Drug: Apatinib Mesylate Tablets

INTERVENTIONS:
Drug: Fluzoparib Capsules — Oral administration of 100 mg, 2 capsules/time (50 mg/capsule), twice daily
Drug: Apatinib Mesylate Tablets — Oral administration of 250 mg each time, 1 tablet/time (250 mg/tablet)

SUMMARY:
Thirty-seven women aged 18-75 years with recurrent ovarian cancer were enrolled

DETAILED DESCRIPTION:
The subjects selected surgery according to the actual situation, and received chemotherapy containing platinum after surgery, totaling 4 cycles of chemotherapy. After the completion of the treatment course, the researchers will use fluzoparil combined with apatinib to maintain the treatment until the disease progression in patients with CR, PR and SD evaluated according to RECIST 1.1 efficacy.

The medication regimen for all enrolled patients was recommended as follows, and the dose could be adjusted during treatment due to adverse reactions and other circumstances:

Fluzopalil capsules:

Oral administration of 100 mg, 2 capsules/time (50 mg/capsule), twice a day, in the morning and evening, before/after meals can be taken orally, it is recommended to take oral administration in the morning and late 0.5h, continuous administration. Every 4 weeks is a treatment period.

Apatinib tablets:

Oral administration of 250 mg each time, 1 tablet/time (250 mg/tablet), it is recommended to take orally 0.5 h after breakfast, continuous administration. Every 4 weeks is a treatment period.

Treatment will continue until an event occurs that meets the criteria for treatment termination.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 ≤75 years old, female; 2. Pathological (including histological) evidence of ovarian epithelial cancer, fallopian tube cancer or primary peritoneal cancer (ovarian cancer); 3. Received first-line platinum drug chemotherapy in the past, the curative effect during the last treatment with platinum regimen (from the start of treatment to within 1 month after the last administration) was non-PD, and the recurrence/progression (platinum resistance) within 6 months after the end of treatment; Or recurrence or progression (platinum-sensitive) ≥6 months after the end of the last platinum-containing treatment; CR/PR/SD after at least 4 cycles of chemotherapy again; 4. According to RECIST1.1 criteria, the patient had at least one target lesion with measurable diameter (tumor lesion with CT scan length ≥10mm, lymph node lesion with CT scan short diameter ≥15mm, and scanning layer thickness 5mm); 5. ECOG PS 0-1 score; 6. Major organs function normally and meet the following criteria:

  1. The standard of blood routine examination must meet: (no blood transfusion within 14 days)

     1. HB≥100g/L,
     2. WBC≥3×109/L
     3. ANC≥1.5×109/L,
     4. PLT≥100×109/L;
  2. Biochemical examination shall meet the following standards:

     1. BIL ≤1.5 times upper limit of normal value (ULN);
     2. ALT and AST≤2.5×ULN, and ALT and AST≤5×ULN in patients with liver metastasis;
     3. Serum Cr≤1.5×ULN. 7. International Standardized ratio (INR) OR prothrombin time (PT), activated partial thrombin activity time (aPTT)≤1.5 × ULN, unless the patient is receiving anticoagulant therapy, as long as PT or aPTT is within the therapeutic range of the anticoagulant drug intended to be used; 8. No serious heart, lung, liver, kidney disorders; 9. Women of reproductive age must undergo a pregnancy test (serological) within 7 days prior to enrollment, with a negative result, and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last dose of the test drug; 10. The expected overall survival ≥6 months, post-treatment survival ≥3 months; 11. Sign a written informed consent and be able to comply with the visit and related procedures specified in the program.

Exclusion Criteria:

1. Other clinical drug experiments in which other experimental drugs are used at the same time as the study;
2. Other cancer treatments, including but not limited to chemotherapy, radiotherapy, targeted therapy, immunotherapy, microbiological therapy, traditional Chinese medicine therapy and other experimental therapies, were used in conjunction with this study;
3. Patients who are known to be allergic to fluzoparil or to active or inactive components of the drug with a similar chemical structure;
4. Patients who are known to be allergic to Apatinib or to active or inactive components of the drug with a similar chemical structure;
5. Inability to swallow oral medications and any gastrointestinal disorders that may interfere with study drug absorption and metabolism, such as uncontrolled nausea and vomiting, gastrointestinal obstruction, or malabsorption;
6. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, including but not limited to surgery, radiation and/or corticosteroids, or clinical manifestations of spinal cord compression;
7. The subject has had other malignant diseases in the past 3 years, except cutaneous squamous cell carcinoma, basal-like carcinoma, ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix;
8. The patient has a prior or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
9. Recent (within 3 months) occurrence of intestinal obstruction, gastrointestinal perforation;
10. Patients with clinical symptoms or diseases that are not well controlled, such as: (1) NYHA2 or above cardiac dysfunction, (2) unstable angina pectoris, (3) acute myocardial infarction occurred within 1 year, (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, (5) QTc>470ms;
11. Any bleeding event with a severe CTCAE 5.0 rating of 2 or more occurring within 4 weeks prior to the initial trial administration;
12. People with hypertension who are not well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
13. Previous or current idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, institutionalized pneumonia, drug-induced pneumonia, or active pneumonia shown by CT during screening;
14. Patients with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds) who have bleeding tendencies or are receiving thrombolytic or anticoagulant therapy (including but not limited to patients requiring long-term anticoagulant therapy) are allowed to receive low-dose low-molecular weight heparin or oral aspirin prophylactic anticoagulant therapy during the trial;
15. Diagnosis of patients with deep vein thrombosis (except intermuscular vein thrombosis);
16. Patients with a history of hereditary or acquired bleeding or coagulation disorders. There were clinically significant bleeding symptoms or definite bleeding tendencies within 3 months before the first trial, such as gastrointestinal bleeding and hemorrhagic gastric ulcer;
17. Subjects with congenital or acquired immune deficiency (such as HIV infection), or active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA≥500 IU/ml; Hepatitis C reference: HCV antibody positive and HCV copy number > upper limit of normal);
18. The patient received platelet or red blood cell transfusions within four weeks prior to initiation of treatment with the investigational drug;
19. Patients who are pregnant or nursing, or who plan to become pregnant during the study treatment period.
20. According to the researchers' judgment, the subjects have other factors that may lead to the forced termination of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to12 months
  To evaluate the efficacy and safety of fluzoparil combined with apatinib for maintenance after platinum-containing chemotherapy in patients with recurrent ovarian cancer by progression-free survival (PFS).

SECONDARY OUTCOMES:
ORR | up to 12 months
  Objective response rate (ORR) was used to evaluate the efficacy of fluzoparil combined with apatinib for maintenance after platinum-containing chemotherapy in patients with recurrent ovarian cancer
OS | up to 24 months
  To evaluate the efficacy of fluzoparil combined with apatinib for maintenance after platinum-containing chemotherapy in patients with recurrent ovarian cancer by overall survival (OS)